CLINICAL TRIAL: NCT06451250
Title: Providing Evidence-Based Approaches for Caregiver Stress (PEACE) Study
Brief Title: Providing Evidence-Based Approaches for Caregiver Stress Study
Acronym: PEACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00008919; 1K01AG066812-01 (NIH)
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Caregiving Stress; Dementia
MeSH Terms: conditions — Caregiver Burden; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult Day Services (Experimental): Adult Day Service use for family member with dementia
  Interventions: Other: Adult Day Service use for family member with dementia

INTERVENTIONS:
Other: Adult Day Service use for family member with dementia — Self-collection of salivary biomarkers 4 times daily for 5 days, two of those days the family member with dementia has to use adult day services

SUMMARY:
The purpose of this preliminary study is to examine the effects of adult day service use on subjective and physiological measures of stress in 50 Black informal caregivers for individuals with dementia (IWD). The PI of the proposed study has substantial training in primary data collection and complex-survey secondary data analysis, she also has the fundamental knowledge to investigate how sociocultural and behavioral factors can influence psychosocial stress. The proposed study will enroll participants from adult day service (ADS) nationally, to examine the effects of adult day service use on subjective and physiological measures of stress in 50 Black informal caregivers. The proposed study extends the current science on the use of ADS on subjective and physiological stress by 1) examining differential impacts of ADS specifically on subjective measures of stress for Black caregivers, 2) evaluating the impact of ADS use on physiological measures of stress among Black caregivers; and 3) examining the relationship between subjective indicators and physiological processes for Black caregivers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older (male or female)
* Self-identify as Black and/or African American,
* Lives with a family member with a physician diagnosis of Alzheimer's disease or related dementia
* Primary responsibility for care of the family member who has been diagnosed with Alzheimer's disease or related dementia
* Utilize Adult Day Services at least two times a week for family member with Alzheimer's disease or related dementia

Exclusion Criteria:

* Either caregiver of client is in active treatment for a terminal illness or are in hospice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2025-12-19 (Actual); Study Completion 2025-12-19 (Actual)

PRIMARY OUTCOMES:
Caregiver stress as assessed by the Perceived Stress Scale | Baseline
  Perceived Stress Scale scores range from 0 to 40 with higher scores indicating higher perceived stress

SECONDARY OUTCOMES:
Salivary cortisol levels | Over a five day period
  Saliva will be collected into sterile collection tubes and stored in participants' freezers until sampling. the test volume will be 25 µL with a sensitivity range of 0.007-3.0 µL/dl.
Salivary alpha-amylase | Over a five day period
  Saliva will be collected into sterile collection tubes and stored in participants' freezers until sampling. the test volume will be 10 µL with a sensitivity range of 0.4-400 U/mL.
Salivary Telomere length | Over a five day period
  Saliva will be collected into sterile collection tubes and stored in participants' freezers until sampling. the test volume will be 2ml

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Parker, PhD, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No